CLINICAL TRIAL: NCT07291869
Title: A Randomised Feasibility Study of Real-time Intracavity ECG and Thoracic Ultrasound for Central Venous Catheter Tip Confirmation in Critical Care
Brief Title: Central Venous Catheter Placement With Thoracic Ultrasound and Intracavity ECG Positioning
Acronym: CVC-TIP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: York Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 360875; 360875 (Other: IRAS)
Record Dates: First submitted 2025-11-21; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Central Venous Catheter; Point of Care Ultrasound (POCUS); Intracavitary Electrocardiogram Guiding; Feasibility Studies
Keywords: Intracavity ECG; POCUS; IC-ECG; Thoracic point of care ultrasound

STUDY DESIGN:
Intervention Model Description: Pragmatic, single-centre, open, randomised control study
Who Masked: Outcomes Assessor
Masking Description: Investigators analysing post-procedure chest x-rays will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LEFT internal jugular vein CVC with IC-ECG and thoracic POCUS (Active Comparator): LEFT internal jugular vein CVC with IC-ECG and thoracic POCUS. Post procedure chest x-ray.
  Interventions: Device: Intracavity ECG; Diagnostic Test: Thoracic point of care ultrasound
- RIGHT internal jugular vein CVC with IC-ECG and thoracic POCUS (Active Comparator): RIGHT internal jugular vein CVC with IC-ECG and thoracic POCUS. Post procedure chest x-ray.
  Interventions: Device: Intracavity ECG; Diagnostic Test: Thoracic point of care ultrasound
- Standard care (No Intervention): Left or right internal jugular vein CVC. Post procedure CXR.

INTERVENTIONS:
Device: Intracavity ECG — Vygon PILOT TLS (Tip Location System) used to provide intracavity ECG monitoring for central venous catheter tip positioning.
  Other Names: IC-ECG
  Arms: LEFT internal jugular vein CVC with IC-ECG and thoracic POCUS; RIGHT internal jugular vein CVC with IC-ECG and thoracic POCUS
Diagnostic Test: Thoracic point of care ultrasound — Thoracic point of care ultrasound used to scan both lung fields to rule out pneumothorax
  Other Names: POCUS
  Arms: LEFT internal jugular vein CVC with IC-ECG and thoracic POCUS; RIGHT internal jugular vein CVC with IC-ECG and thoracic POCUS

SUMMARY:
The goal of this interventional study is to assess the feasibility of two bedside techniques for confirming central venous catheter (CVC) placement and detecting complications:

* Intracavity ECG monitoring to confirm internal jugular vein CVC tip position.
* Thoracic point-of-care ultrasound (POCUS) to rule out pneumothorax following CVC insertion.

Participants who require an internal jugular CVC as part of their routine care and meet all inclusion and no exclusion criteria will be randomised to receive either:

* Standard care, or
* The intervention, consisting of intracavity ECG guidance and thoracic POCUS. The CVC will be inserted either on the left or right side of the neck.

All participants will undergo a post-procedure chest X-ray regardless of study arm, to allow comparison of the intervention methods with standard care.

DETAILED DESCRIPTION:
Central venous catheters (CVCs) are commonly inserted in critically ill patients to enable the administration of medications, fluids, and monitoring. Following insertion, it is standard practice to perform a chest X-ray (CXR) to confirm correct catheter tip position and exclude complications such as pneumothorax. However, reliance on post-procedure radiography can delay verification of line position, increase patient radiation exposure, and contribute to workflow inefficiency.

Alternative bedside techniques have been proposed to improve the speed and safety of CVC verification. Intracavity electrocardiography (IC-ECG) uses the patient's cardiac electrical activity to confirm the catheter tip's location in real time. When the catheter tip approaches the cavoatrial junction, a characteristic increase in P-wave amplitude is observed, allowing for accurate placement without the need for immediate imaging. Thoracic point-of-care ultrasound (POCUS) has been shown to be an effective method for detecting pneumothorax following CVC insertion.

This single-centre, prospective, randomised feasibility study will evaluate the combined use of intracavity ECG for tip confirmation and thoracic POCUS for pneumothorax exclusion in patients requiring internal jugular CVC insertion. Eligible participants will be randomised to receive either:

* Standard care (ultrasound-guided insertion with post-procedure CXR), or
* The intervention, consisting of ultrasound-guided insertion supplemented with intracavity ECG confirmation and thoracic POCUS assessment, followed by a post-procedure CXR for comparison.

The primary objective is to determine the feasibility of implementing these combined techniques within a critical care environment, including assessment of recruitment, protocol adherence, and completeness of data acquisition. Secondary outcomes include the accuracy of IC-ECG and POCUS compared to CXR for tip position and pneumothorax detection, and the time required to confirm line placement.

The findings will inform the design of a future multi-centre study to assess diagnostic accuracy, cost-effectiveness, and potential to replace routine post-procedure chest X-ray in appropriate clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged ≥ 18 years)
* Admitted, or planned for admission, to critical care
* Requiring central venous catheter insertion as a part of their usual care
* Suitable for both right or left internal jugular vein insertion

Exclusion Criteria:

* Previously randomised into CVC-TIP
* Atrial fibrillation on 12-lead ECG
* Cardiovascular instability, defined as
* Noradrenaline dose > 0.5mcg/kg/min
* Rapidly escalating doses of vasopressors / inotropes
* Difficulty in obtaining thoracic ultrasound images due to either
* Weight > 120kg
* Existing pneumothorax (either side)
* Subcutaneous emphysema
* Wounds / dressing over anterior chest wall
* Existing pacemaker
* Non-English speaking participants
* Death perceived as imminent
* Any other reason as determined by treating clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | 12-month recruitment window
  How quickly the recruitment target can be achieved within the planned study period
Protocol adherence | 12-month recruitment window
  The number of protocol deviations for all 3 arms
Data completeness | 12-month recruitment window
  The percentage complete data records for each enrolment
Training requirements | 12-month recruitment window
  Feasibility of delivering the required clinician training to ensure safe and consistent implementation of the study protocol
Technical success rate | 12-month recruitment window
  How successful the intervention is when compared to the gold standard chest x-ray
Time taken for confirmation of central venous catheter tip positioning | 12-month recruitment window
  Time taken from start of procedure to successful confirmation (both using intracavity ECG and chest x-ray)

SECONDARY OUTCOMES:
Rate of catheter malposition | 12-month recruitment window
  The incidence of central venous catheter malposition on intracavity-ECG and chest x-ray in all treatment arms
Incidence of complications | Insertion to 48 hours post-procedure
  Rate of procedure-related complications occurring during or immediately after insertion.
Inter-operator reliability of IC-ECG and POCUS findings | Images stored during the procedure and reviewed up to 28 days post-procedure
  Measurement of inter-operator reliability for IC-ECG and POCUS interpretations, using blinded independent review of stored image and waveform data.
Proportion of cases which would avoid post-insertion CXR | 12-month recruitment window
  Proportion of catheter insertions where post-procedural a chest x-ray would not be required based on the study criteria
Operator confidence | Completed within 24 hours of catheter insertion
  Operator survey for each procedure in the intervention arm, which includes a 5-point Likert confidence scale from "Not Confident" to "Extremely Confident"

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Chamberlain, MBChB, Principal Investigator — York Teaching Hospitals NHS Foundation Trust
Locations (1):
- York and Scarborough Teaching Hospitals NHS Foundation Trust, York, North Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised individual participant data will not be publicly available. Data may be shared on reasonable request with approval from the trial steering committee and subject to a signed data sharing agreement. Shared data will include de-identified procedural and clinical outcome information and may be used for secondary analyses or meta-analyses.

REFERENCES:
- [Background] Fletcher SJ, Bodenham AR. Safe placement of central venous catheters: where should the tip of the catheter lie? Br J Anaesth. 2000 Aug;85(2):188-91. doi: 10.1093/bja/85.2.188. No abstract available. PMID 10992821
- [Background] Kang M, Bae J, Moon S, Chung TN. Chest radiography for simplified evaluation of central venous catheter tip positioning for safe and accurate haemodynamic monitoring: a retrospective observational study. BMJ Open. 2021 Jan 4;11(1):e041101. doi: 10.1136/bmjopen-2020-041101. PMID 33397666